CLINICAL TRIAL: NCT03795649
Title: The Immunomodulatory Effect of Antrifibrinolytic (Tranexamic Acid) in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sisters of Mercy University Hospital (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Renata Letica-Brnadić, Principal Investigator, Sisters of Mercy University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EP-12939/18-1
Record Dates: First submitted 2018-12-30; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The control group (Group K) (No Intervention): The control group (Group K) is comprised of surgical patients who will not receive blood transfusion, and who have contraindications for Tranexamic Acid.
- Group A, Tranexamic acid (Active Comparator): The treatment group (Group A) is comprised of the patients who will receive Tranexamic acid 1g intravenous 15 min. before releasing the pneumatic tourniquet and the repeating dose 3 hours later
  Interventions: Drug: Tranexamic Acid
- Group B, autologous transfusion (Other): The treatment group (Group B) will be comprised of the patients who in the second selection have one or more contraindications for Tranexamic Acid administration and transfusion of autologous blood will be performed.
  Interventions: Drug: Tranexamic Acid
- Group C, alogenous transfusion (Other): The treatment group (Group C) contraindications for Tranexamic Acid administration and the transfusion of alogenous blood will be performed in the case of acute haemorrhage followed by patient's hemodynamic instability.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Imunomodulatory effect
  Other Names: Medsamic
  Arms: Group A, Tranexamic acid; Group B, autologous transfusion; Group C, alogenous transfusion

SUMMARY:
The administration of the tranexamic acid (TRAXA), an antifibrinolytic, blocks primary fibrinolysis, and thus the haemorrhage, in the early postoperative period. Significant surgical operations, as well as trauma, initiate a similar dynamic homeostatic mechanism between the creation of a clot (primary and secondary haemostasis) and its dissolution (fibrinolysis). Antifibrinolytics have been proven effective in reducing haemorrhage in patients who have undergone significant surgical operations with normal fibrinolysis, with the use of an appropriate surgical technique.

A pharmacokinetic study has shown that peak fibrinolytic activity is present for 6 hours after the incision and it persists for 18 hours in total knee and hip arthroplasty. The administration of the tranexamic acid in optional orthopaedic surgery of total hip (THA) and knee (TKA) arthroplasty reduces the postoperative haemorrhage, as well as the number and volume of the postoperative autologous blood.

A trauma in the organism triggers the immunologic response. New term has been introduced - the post-traumatic immunosuppression (PTI), characterised by: a change on the immunologic cells (neutrophilia, monocytosis, increased number of mesenchymal stromal cells, reduced expression of HLA-DR on monocytes, reduced function of natural killer (NK) cells, increased lymphocyte apoptosis, a shift in homoeostasis towards the Th2 phenotype facilitated by Treg lymphocytes - CD4+CD25+CD127-); a change in production levels of various cytokines (anti-inflammatory cytokines): IL-10, IL-4; anti- and pro-inflammatory cytokine: IL-6; pro-inflammatory cytokines IL-2, TNF-α, IFN-γ); the activation of the complement system (C5a and C3a via factor VII - tissue factor system, activated by cell damage).

Post-traumatic immunosuppression can be made worse by transfusion, haemorrhage, stress, significant surgical operation and immunosuppressive drugs.

The research has shown that Treg lymphocytes CD4+CD25+CD127- have an important role in controlling the acquired and innate immunity (comprising 6-8% of all CD4+ lymphocytes).

Stopping haemorrhage prevents the occurrence of anaemia, as well as the need for transfusion of blood products, which lead to developing the post-traumatic immunosuppression (PTI).

DETAILED DESCRIPTION:
The administration of the tranexamic acid (TRAXA), an antifibrinolytic, blocks primary fibrinolysis, and thus the haemorrhage, in the early postoperative period. Significant surgical operations, as well as trauma, initiate a similar dynamic homeostatic mechanism between the creation of a clot (primary and secondary haemostasis) and its dissolution (fibrinolysis). Antifibrinolytics are initially used in patients with an accelerated fibrinolysis of different pathogeneses. However, they have been proven effective in reducing haemorrhage in patients who have undergone significant surgical operations with normal fibrinolysis, with the use of an appropriate surgical technique.

A pharmacokinetic study has shown that peak fibrinolytic activity is present for 6 hours after the incision and it persists for 18 hours in total knee and hip arthroplasty. The administration of the tranexamic acid in optional orthopaedic surgery of total hip (THA) and knee (TKA) arthroplasty reduces the postoperative haemorrhage, as well as the number and volume of the postoperative autologous blood.

A randomized, placebo-controlled trial CRAS-2 has validated that the early post-traumatic administration of the tranexamic acid, within 8 hours after the injury, in adult patients with traumas or in patients with the risk of significant haemorrhage, reduces the fatality rate.

The tranexamic acid is a synthetic derivative of lysine, an amino acid which blocks lysine binding sites of the plasminogen molecule which are essential for its biding to fibrin. This mechanism inhibits the plasminogen activation via a plasminogen activator which also binds to fibrin. Thus, it prevents the conversion of plasminogen into plasmin, which is essential for fibrin dissolution, the integral element of a stable clot. The second important antifibrinolytic effect is blocking the lysine binding sites on the free plasmin molecule which has already been formed through the conversion from the plasminogen. This inhibits its binding to fibrin, and the TRAXA-plasmin complex is rapidly inactivated with the α-2-antiplasmin and α-2-macroglobulin. Biological half-life is approximately 2-3 hours.

A trauma in the organism triggers the immunologic response. The initial immunologic reaction occurs at the location of the injury, and it is called an inflammation. The inflammatory response is characterized by a complex interaction of macrophages (a type of leukocytes which develop from monocytes and are a part of the mononuclear phagocyte system, the main task of which are phagocytosis, i.e. the clearance of foreign materiel from the organism, performing the immunologic function - the defence against foreign materiel - antigens, and the regulation of the inflammation via interleukins which they secrete - IL1, IL-2,TNF) and dendritic cells (antigen-presenting cells), the consequence of which is the release of cytokines (interleukins - glycoproteins which regulate interactions among cells) and chemokine (small proteins from the cytokine group - able to induce chemotaxis, cell migration), and the activation of the neutrophils, monocytes and mesenchymal stem cells (cells not containing any information, located in the adipose tissue, cartilage and muscle tissue).

If the initial inflammatory response at the location of the injury is strong enough, it will develop into a systemic inflammatory response, called systemic inflammatory response syndrome (SIRS), which implies an inflammatory response of the entire body without a proven source of infection. The criteria for the diagnosis of the SIRS are: heart rate higher than 90 bpm; body temperature lower than 36°C or higher than 38°C; tachypnoea, respiratory rate higher than 20 breaths per minute or the partial pressure of carbon dioxide in the blood lower than 4.3 kPa (32 mm Hg); the number of white blood cells, leukocytes, lower than 4.000 cells in 1 mm³ or higher than 12.000 cells in 1 mm³; or the presence of more than 10% of immature neutrophils. A destructive immunologic inflammatory cascade can prevent or delay healing.

At the same time the compensatory anti-inflammatory response syndrome (CARS) is initiated, which includes the immunologic response with the aim of re-establishing the immunologic homeostasis. It is characterized by: a reduced cytokine response of monocytes to the stimulation; a reduced number of antigen-presenting receptors (human leukocyte antigens or HLA) on monocytes; an increased level of IL-10, an anti-inflammatory cytokine; lymphocyte apoptosis (T-cells); lymphocyte dysfunction, i.e. reduced proliferation; reduced Th1 proinflammatory cytokine production (a shift in homoeostasis towards the Th2 phenotype facilitated by the regulatory T lymphocytes). It clinically manifests as skin allergy, hypothermia and leukopenia. Additional criteria include elevated levels of C-reactive proteins, lactates and hyperglycaemia. If the immunosuppressive response persists, it may increase the possibility of an infection occurring, and the inability to defend against the infection, which may result in the development of sepsis, multiple organ failure and death.

Due to the wide clinical and laboratory criteria which both the SIRS and CARS terms include, they are not the best terms for describing the immunologic response to a trauma, and a new term has been introduced - the post-traumatic immunosuppression (PTI), characterised by: a change on the immunologic cells (neutrophilia, monocytosis, increased number of mesenchymal stromal cells, reduced expression of HLA-DR on monocytes, reduced function of natural killer (NK) cells, increased lymphocyte apoptosis, a shift in homoeostasis towards the Th2 phenotype facilitated by Treg lymphocytes - CD4+CD25+CD127-); a change in production levels of various cytokines (anti-inflammatory cytokines): IL-10, IL-4; anti- and pro-inflammatory cytokine: IL-6; pro-inflammatory cytokines IL-2, TNF-α, IFN-γ); the activation of the complement system (C5a and C3a via factor VII - tissue factor system, activated by cell damage).

Post-traumatic immunosuppression can be made worse by transfusion, haemorrhage, stress, significant surgical operation and immunosuppressive drugs.

The research has shown that Treg lymphocytes CD4+CD25+CD127- have an important role in controlling the acquired and innate immunity (comprising 6-8% of all CD4+ lymphocytes).

The normal function of Treg lymphocytes is the suppression of the T-cell response against its own antigens.

Stopping haemorrhage prevents the occurrence of anaemia, as well as the need for transfusion of blood products, which lead to developing the post-traumatic immunosuppression (PTI).

Monitoring the immunologic status of patients with the understanding of the PTI mechanism can enable timely and individual modulation of the immunologic status with pre-planned procedures (preventing haemorrhage, anaemia, avoiding transfusion) and/or immunotherapy (drugs and nutrients), and thereby prevent the occurrence of complications, such as infections. Infections may result in sepsis and multiple-organ failure, and eventually be lethal for the patient.

The research has proved that Treg lymphocytes CD4+CD25+CD127- have an important role in controlling the acquired and innate immunity (comprising 6-8% of all CD4+ lymphocytes).

The normal function of Treg lymphocytes is the suppression of the T-cell response against its own antigens.

There are two main types of regulatory lymphocytes: natural Treg, which are mostly developed in the thymus, and inducible Treg, which arise in the periphery after being exposed to cytokines, antigen-presenting cells or immunosuppressive drugs. It may be difficult to differentiate these two lymphocyte Treg populations in vivo. Nevertheless, it is known that different stages of the infection require different regulations. Acute infection, tissue damage, inflammation caused by the innate immunologic response is limited, i.e. locally controlled via natural Treg lymphocytes. This mechanism triggers the activation of inducible Treg lymphocytes.

For the first time, in 1995, it was described that the suppression of CD4+ T-lymphocytes is caused by a low T-cell population with the CD4+ CD25+ expression. Natural Treg lymphocytes, apart from belonging to CD4+ T-cell population, have a CD25+ receptor, an α-receptor chain for IL-2, and a receptor for the cytotoxic T-lymphocytic antigen 4 (CTLA 4), the tumour necrosis factor receptor (TNF), but it differs from the activated T-cells by the expression of the transcription factor FoxP3 (transcription factor encoded with the FoxP3 gene). The expression of CD 127lo, an α-chain receptor for the interleukin 7 enables us to differentiate Treg lymphocytes from the activated T-lymphocytes via flow cytometry. The number of CD25+CD127lo cells correlates to the number of CD25+FoxP3+ cells in the peripheral blood.

Different studies show that the application of the 3-colour flow cytometry shows small variation in the percentage of Treg lymphocytes in the peripheral blood from 6.35% to 8.34%.

There is a number of different mechanisms which achieve regulation by using the Treg lymphocytes: the long-term interaction with dendritic cells (DC), thereby modulating the function of antigen-presenting cells (APC), the production of the anti-inflammatory cytokine, IL-10 and the CTLA4 expression on Treg cells which induces the enzyme indoleamine 2,3-dioxygenase (IDO) in APC which degrade the amino acid tryptophan, the lack of which inhibits the activation of T-cells and induces T-cell apoptosis. Treg lymphocytes also induce the apoptosis of monocytes and affect the lower expression of HLA-DR on monocytes whereby they directly affect the innate immunological response.

Elevated, suppressive activity of Treg cells in traumas prevents the protective Th1 response for up to 7 days in comparison with the healthy population.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II status
* scheduled for endoprosthetic total knee arthroplasty.
* laboratory results suitable for elective endoprosthetic surgery: blood panel, coagulation, liver enzymes, kidney function parameters, urine sediment;
* patient voluntarily, in accordance with the KBCSM form on the administration of Tranexamic Acid in endoprosthetic total knee arthroplasty, give their consent for its administration.
* signed informed consent for transfusion

Exclusion criteria:

* general anaesthesia
* revision arthroplasty
* previous blood transfusions
* known allergic reaction to TRAXA
* presence of an infection and/or acutization of a chronic disease
* existing malignant disease
* autoimmune disease
* hematologic disease
* diabetes
* renal failure
* liver cirrhosis
* chronic anticoagulant therapy
* analgesia by non-steroidal anti-inflammatory drugs
* combined use of the autologous and allogeneic blood postoperatively when the recovery of the autologous blood is insufficient in relation to the haemorrhage.

Exclusion Criteria refers to the patients for whom Tranexamic Acid was contraindicated: ----thromboembolic events (IM, CVI, DVT)

* known risk of thrombosis or thromboembolic events (thrombogenic valve disease, thrombogenic rhythm disorder, coagulation-hypercoagulation disorder)
* epilepsy
* patients who use oral contraceptives
* known retinal arterial or venous occlusions.

To patients who fulfil the participation criteria for the trial in the first selection, and for whom TRAXA is contraindicated in the second selection, blood transfusion will be administered in accordance with the indication.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The immunomodulation effect of Tranexamic Acid (IM) | two years
  Trial will include approximately 100 patients in total, which will be divided into four groups of 25 patients. The immunomodulation effect is monitored through the analysis of the lymphocyte subpopulation in the peripheral blood through flow cytometry.
  The result of each lymphocyte subpopulation will be registered as a percentage of all helper cells (CD4+) and all lymphocytes, as well as their absolute number in the peripheral blood.
  These parameters will be monitored dynamically in the chronological order as shown below:
  Day 1 - Preoperatively; Day 1 - Postoperatively T1 (IM) K - 6 hrs postoperatively T1 (IM) A - 6 hrs after the first TRAXA dose, and two hours before LMWH T1 (IM) B - 6 hrs postoperatively (after the transfusion of the autologous blood by means of the autotransfusion system); Day 3 - Postoperatively; Day 5 - Postoperatively; Day 7 - Postoperatively; For immunologic testing of each patient's blood 25 ml (5 ml x 5) during 7 days will be sampled.

SECONDARY OUTCOMES:
The effect of the Tranexamic Acid on the primary fibrinolysis (F) | two years
  The fibrinolytic activity of plasma will be examined through euglobulin lysis time testing Blood sampling follows the same time intervals of blood sampling for determining Treg lymphocytes. Fibrinolysis is monitored until the third postoperative day.
  In total per patient for analysis of the fibrinolytic activity 15 mL (5 mL x 3) of blood will be sampled during a 3-day period.
  Day 1 - Preoperatively; Day 3 - Postoperatively T1 (F) K - 6 hrs postoperatively T1 (F) A - 6 hrs after the first TRAXA dose, and two hours before LMWH T1 (F) B - 6 hrs postoperatively (after the transfusion of the autologous blood by means of the autotransfusion system); Day 3 - Postoperatively;

CONTACTS AND LOCATIONS:
Overall Officials: Renata Letica-Brnadić, Study Chair — Clinical Hospital Centre "Sisters of Mercy"
Locations (1):
- Klinički Bolnički Centar Sestre Milosrdnice, Zagreb, Croatia

REFERENCES:
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, McClelland B, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001886. doi: 10.1002/14651858.CD001886.pub2. PMID 17943760
- [Background] Astedt B. Clinical pharmacology of tranexamic acid. Scand J Gastroenterol Suppl. 1987;137:22-5. PMID 3321402
- [Background] Roberts I, Shakur H, Coats T, Hunt B, Balogun E, Barnetson L, Cook L, Kawahara T, Perel P, Prieto-Merino D, Ramos M, Cairns J, Guerriero C. The CRASH-2 trial: a randomised controlled trial and economic evaluation of the effects of tranexamic acid on death, vascular occlusive events and transfusion requirement in bleeding trauma patients. Health Technol Assess. 2013 Mar;17(10):1-79. doi: 10.3310/hta17100. PMID 23477634
- [Background] Oremus K, Sostaric S, Trkulja V, Haspl M. Influence of tranexamic acid on postoperative autologous blood retransfusion in primary total hip and knee arthroplasty: a randomized controlled trial. Transfusion. 2014 Jan;54(1):31-41. doi: 10.1111/trf.12224. Epub 2013 Apr 25. PMID 23614539
- [Background] Raveendran R, Wong J. Tranexamic acid: more evidence for its use in joint replacement surgery. Transfusion. 2014 Jan;54(1):2-3. doi: 10.1111/trf.12494. No abstract available. PMID 24405302
- [Background] Parkin J, Cohen B. An overview of the immune system. Lancet. 2001 Jun 2;357(9270):1777-89. doi: 10.1016/S0140-6736(00)04904-7. PMID 11403834
- [Background] Islam MN, Bradley BA, Ceredig R. Sterile post-traumatic immunosuppression. Clin Transl Immunology. 2016 Apr 29;5(4):e77. doi: 10.1038/cti.2016.13. eCollection 2016 Apr. PMID 27195120
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Bone RC. Immunologic dissonance: a continuing evolution in our understanding of the systemic inflammatory response syndrome (SIRS) and the multiple organ dysfunction syndrome (MODS). Ann Intern Med. 1996 Oct 15;125(8):680-7. doi: 10.7326/0003-4819-125-8-199610150-00009. PMID 8849154
- [Background] Ward NS, Casserly B, Ayala A. The compensatory anti-inflammatory response syndrome (CARS) in critically ill patients. Clin Chest Med. 2008 Dec;29(4):617-25, viii. doi: 10.1016/j.ccm.2008.06.010. PMID 18954697
- [Background] Osuka A, Ogura H, Ueyama M, Shimazu T, Lederer JA. Immune response to traumatic injury: harmony and discordance of immune system homeostasis. Acute Med Surg. 2014 Jan 28;1(2):63-69. doi: 10.1002/ams2.17. eCollection 2014 Apr. PMID 29930824
- [Background] Seddiki N, Santner-Nanan B, Martinson J, Zaunders J, Sasson S, Landay A, Solomon M, Selby W, Alexander SI, Nanan R, Kelleher A, Fazekas de St Groth B. Expression of interleukin (IL)-2 and IL-7 receptors discriminates between human regulatory and activated T cells. J Exp Med. 2006 Jul 10;203(7):1693-700. doi: 10.1084/jem.20060468. Epub 2006 Jul 3. PMID 16818676
- [Background] Venet F, Chung CS, Kherouf H, Geeraert A, Malcus C, Poitevin F, Bohe J, Lepape A, Ayala A, Monneret G. Increased circulating regulatory T cells (CD4(+)CD25 (+)CD127 (-)) contribute to lymphocyte anergy in septic shock patients. Intensive Care Med. 2009 Apr;35(4):678-86. doi: 10.1007/s00134-008-1337-8. Epub 2008 Oct 23. PMID 18946659
- [Background] Venet F, Chung CS, Monneret G, Huang X, Horner B, Garber M, Ayala A. Regulatory T cell populations in sepsis and trauma. J Leukoc Biol. 2008 Mar;83(3):523-35. doi: 10.1189/jlb.0607371. Epub 2007 Oct 3. PMID 17913974
- [Background] Belkaid Y. Regulatory T cells and infection: a dangerous necessity. Nat Rev Immunol. 2007 Nov;7(11):875-88. doi: 10.1038/nri2189. PMID 17948021
- [Background] Shevach EM, DiPaolo RA, Andersson J, Zhao DM, Stephens GL, Thornton AM. The lifestyle of naturally occurring CD4+ CD25+ Foxp3+ regulatory T cells. Immunol Rev. 2006 Aug;212:60-73. doi: 10.1111/j.0105-2896.2006.00415.x. PMID 16903906
- [Background] Hartigan-O'Connor DJ, Poon C, Sinclair E, McCune JM. Human CD4+ regulatory T cells express lower levels of the IL-7 receptor alpha chain (CD127), allowing consistent identification and sorting of live cells. J Immunol Methods. 2007 Jan 30;319(1-2):41-52. doi: 10.1016/j.jim.2006.10.008. Epub 2006 Nov 3. PMID 17173927
- [Background] Fragkou PC, Torrance HD, Pearse RM, Ackland GL, Prowle JR, Owen HC, Hinds CJ, O'Dwyer MJ. Perioperative blood transfusion is associated with a gene transcription profile characteristic of immunosuppression: a prospective cohort study. Crit Care. 2014 Oct 1;18(5):541. doi: 10.1186/s13054-014-0541-x. PMID 25270110
- [Result] Blanie A, Bellamy L, Rhayem Y, Flaujac C, Samama CM, Fontenay M, Rosencher N. Duration of postoperative fibrinolysis after total hip or knee replacement: a laboratory follow-up study. Thromb Res. 2013 Jan;131(1):e6-e11. doi: 10.1016/j.thromres.2012.11.006. Epub 2012 Nov 26. PMID 23195143